CLINICAL TRIAL: NCT02878187
Title: Evaluation of the Uterine Cavity and Blood Flow After Conservative Management of Placenta Previa/Accreta
Brief Title: Uterine Cavity and Blood Flow After Conservative Management of Placenta Previa/Accreta
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Other Study IDs: PP
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Improving Quality of Life
MeSH Terms: interventions — Echocardiography, Doppler

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- placenta previa: all women managed by conservative surgical techniques during cesarean section after intraoperative hemorrhage due to placenta previa/accreta
  Interventions: Device: Doppler
- healthy controls: women delivered by Cesarean for any other indication with no intraoperative hemorrhage or any additional surgical techniques performed during Cesarean
  Interventions: Device: Doppler

INTERVENTIONS:
Device: Doppler — Color Doppler ultrasound will be used to demonstrate the main ascending branches of left and right uterine arteries as they cross over the hypogastric vessels just before they enter the uterus at the uterine-cervical junction. The high pass filter was set at 125 Hz and the uterine artery will be obtained immediately after the crossing of the hypogastric artery. The sample volume will be placed on the artery with an angle of about 0°. After detection of blood flow and visu¬alization of the waveform of the uterine artery, five blood flow indices will be automatically cal¬culated:
  The pulsatility index The resistance index The peak systolic velocity ; The end-diastolic velocity The time-averaged maximum

SUMMARY:
Bleeding is the most significant cause of maternal death worldwide with more than half of those occurring within the first day of delivery. About 10.5% (some estimate as high at 12-17%) of live births world-wide, or about 14 million births, are complicated by postpartum hemorrhage; a woman dies every 4 minutes from postpartum hemorrhage. Uterine atony and placenta accreta are the two leading causes of postpartum hysterectomies with up to 64% of Cesarean hysterectomies done for abnormally adherent placentation

DETAILED DESCRIPTION:
No previous studies performed for evaluation of the effect of those procedures on the uterine cavity or uterine blood flow. Most of the studies in the literature evaluated the menstrual and fertility outcome after conservative measures for intraoperative hemorrhage due to placenta previa/accreta were retrospective and depend on the resumption of menses and pregnancy rate

ELIGIBILITY:
Inclusion Criteria:

1. Women Age 18-40 years
2. Gestational age of pregnancy 28-40 weeks
3. Diagnosed antenatally as placenta previa/accreta
4. Patients who will be managed by conservative surgical techniques for intraoperative hemorrhage
5. Women who will accept to participate in the study and are reliable for follow-up

Exclusion Criteria:

* 1- Patients who will be managed by hysterectomy 2- Patients who will be managed by conservative leaving the placenta in-situ 3- Diabetic or hypertensive women 4- Women who will refuse to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women delivered by elective/emergency cesarean section due to placenta previa/accreta during the study period will be included in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
The mean difference in the uterine arteries diameters in both groups | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abbas, MD, Principal Investigator — Assiut University
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes